CLINICAL TRIAL: NCT05358808
Title: ACHIEVE - An Adaptive Trial of the Efficacy and Effectiveness of Adoptive Cellular tHerapy wIth Ex-Vivo Expanded Allogeneic γδ T-lymphocytes (TCB008) for Patients With Refractory or Relapsed Acute Myeloid Leukaemia (AML)
Brief Title: ACHIEVE - Efficacy and Effectiveness of Adoptive Cellular tHerapy wIth Ex-Vivo Expanded Allogeneic γδ T-lymphocytes (TCB008) for Patients With Refractory or Relapsed Acute Myeloid Leukaemia (AML)
Acronym: ACHIEVE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Trial was early terminated due to deficiencies in the Achieve Protocol: V8.0 dated 19 January 2024.
Sponsor: TC Biopharm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCB008-001
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
Keywords: AML; MDS; MDS/AML; AML/MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Receptors, Antigen, T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- γδ T cells (IMP, TCB008) (Experimental): After inclusion, all patients will receive lymphodepleting chemotherapy with fludarabine 30mg/m2 Day -6 to Day -3 [total 120 mg/m2] and cyclophosphamide 0.5g/m2 [total 1.5 g/m2) Day -5 to Day -3,]. This will be followed by a rest day (Day -2).
  The first five patients (safety cohort) will receive 1.8mL of TCB008 (containing 3.5x10^7 to 11.0x10^7 cells) on Day 0.
  After treatment of the first five safety patients, the remaining 48 patients will receive 5mL of TCB008 (containing 12.0x10^7 to 23.0x10^7 cells) on Day 0.
  Interventions: Drug: TCB008

INTERVENTIONS:
Drug: TCB008 — TCB008 is derived from the peripheral blood mononuclear cells (PBMCs) of unrelated, healthy donors and consists of expanded cluster designation (CD)3+ T cells expressing the γ chain variable region 9 δ-chain variable region 2 (Vγ9Vδ2) T cell receptor (TCR); it is infused into patients to boost their immune system. It is currently developed for treatment of cancers and infectious diseases.
  Other Names: CD3+ T cells expressing the γ-chain variable region 9 δ-chain variable region 2 (Vγ9Vδ2) T cell receptor (TCR)

SUMMARY:
This is an open-label, phase II study designed to evaluate the efficacy and effectiveness of TCB008 in patients with Acute Myeloid Leukemia (AML), or Myelodysplastic Syndromes (MDS)/AML, with either refractory or relapsed disease.

Five patients will be recruited for an initial safety cohort. The safety cohort will be followed by a two-stage Simon's Design, where a further 48 patients will be recruited into one of two cohorts and dosed with TCB008.

DETAILED DESCRIPTION:
TCB008-001 (ACHIEVE) is an open-label, phase II study designed to evaluate the efficacy and effectiveness of TCB008 in patients with Acute Myeloid Leukemia (AML), or Myelodysplastic Syndromes (MDS)/AML, with either refractory or relapsed disease.

TCB008 is derived from the peripheral blood mononuclear cells (PBMCs) of unrelated, healthy donors and consists of expanded cluster designation (CD)3+ T cells expressing the γ-chain variable region 9 δ-chain variable region 2 (Vγ9Vδ2) T cell receptor (TCR); it is infused into patients to boost their immune system. It is currently developed for treatment of cancers and infectious diseases.

53 patients will take part in this study; five patients in an initial safety cohort followed by a two-stage Simon's Design that will recruit a further 48 patients into one of two patient cohorts.

Patients will be screened to assess their eligibility to enter the study 35 days prior to the first dose of the investigational medicinal product (IMP). Once enrolled in the study, patients will undergo lymphodepletion chemotherapy prior to administration of the IMP using the following regimen: fludarabine (30mg/m2/day) will be administered from days -6 to -3 (total 120mg/m2), and cyclophosphamide (0.5g/m2/day) from days -5 to -3 (total 1.5g/m2). No chemotherapy will be administered on days -2 and -1.

Cohort A will recruit patients with relapsed or refractory AML or MDS/AML. These patients will be split between one of two sub-cohorts;

* Cohort A1 will include patients with primary refractory AML or MDS/AML who have not achieved a CR, CRi, or CRh after two cycles of induction chemotherapy.
* Cohort A2 will include patients with AML or MDS/AML who have relapsed after initially achieving a CR, CRi, or CRh to previous chemotherapy.

This cohort would include MDS/AML patients with 10 to 19% blast levels in the bone marrow or peripheral blood as defined in the European Leukemia Net 2022 Criteria (as per international consensus classification of AML).

Cohort B will recruit patients with AML or MDS/AML who have achieved CR, CRi, or CRh but have a detectable measurable residual disease by MFC-MFD or Mol-RD by qPCR.

Patients may receive repeat infusions of TCB008, on up to three occasions, 14 days after the previous infusion. Re-infusions will not be preceded by lymphodepleting chemotherapy.

Patients will be followed for up to 52 weeks following the first infusion of TCB008, or until either; they are lost to follow-up, or early termination. Blood and bone marrow samples will be taken pre- and post-infusion to evaluate the study objectives and endpoints.

The total duration of study participation for each patient, from screening through to the end of study visit, is anticipated to be approximately 15 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 at the time of consent
2. Karnofsky performance status ≥ 70% and WHO/ECOG performance status 0 -1 at enrolment and up to 2 at the time of infusion.
3. Must be able to remain free of systemic corticosteroid (e.g., prednisolone) and other immunosuppressive therapy at screening and for at least 5 days prior to the infusion of γδ T cells. Maintenance replacement steroid after assessment of the primary endpoint is permitted.
4. Must be able to understand and sign written informed consent and willing to participate in a clinical trial for an advanced therapy investigational medicinal product (AT(I)MP).
5. For women of childbearing potential, a urine or serum pregnancy test will be performed within 7 days prior to initiating lymphodepletion. A serum pregnancy test will be performed on the day prior to the first infusion of TCB008 (i.e. day -1) and urine or serum pregnancy tests will be performed on the day of subsequent infusions with TCB008 and the results must be negative at all times that these pregnancy tests are performed. For women of childbearing potential, a serum pregnancy test will be performed at visit 17 or early termination. Patient and his/her partner must agree to use adequate contraception from the time of providing written consent through 3 months after the last study drug dose
6. Pathologically confirmed diagnosis of AML or MDS/AML confirmed according to ELN 2022 Criteria (as per International Consensus Classification of AML).
7. For Cohort A1, patients must have AML or MDS/AML that is primary refractory defined as not achieving a CR, CRi or CRh after 2 cycles of intensive or non-intensive induction chemotherapy.
8. For Cohort A2, patients with AML or MDS/AML must have previously achieved a CR, CRi or CRh (including MRD negative CR) to previous intensive or non-intensive therapy, then have experienced relapsed AML.
9. For Cohort B, patients with AML who have achieved CR, CRi or CRh but have persistent MRD by multiparameter flow cytometry-based MRD (MFC-MRD) or molecular MRD (Mol-MRD) assessed by qPCR.

Included patients will not be deprived of standard of care by participating in this trial.

Exclusion criteria

1. Suspected or proven active CNS disease.
2. Previous reactions to Fludarabine or Cyclophosphamide or patients at risk of Fludarabine related neurotoxicity
3. Acute promyelocytic leukaemia
4. Bisphosphonates (≤8 weeks before study entry), unless continued as a standard of care medication
5. Corticosteroids (cumulative dose of systemic steroids >20mg of prednisolone per day or equivalent) that cannot be discontinued 5 days prior to TCB008 infusion.
6. Antihyperlipidemic medications (e.g., statins) that cannot be discontinued prior to enrolment.
7. Cardiac failure: EF < 40%.
8. Kidney function: creatinine clearance ≤ 60 mL/min.
9. Liver function: total bilirubin > 3 × ULN, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) > 5 × ULN.
10. Neurological condition(s) which might be exacerbated by therapy or prevent assessments for neurotoxicity/ICANS.
11. GVHD of any grade or anti-GVHD treatment.
12. Lung function: symptoms of respiratory failure or < 92% oxygen saturation on air.
13. Active infections that are difficult to control, including positive COVID-19 diagnosis at screening. NOTE: Active infections following lymphodepletion may exclude a patient from being able to be dosed with IMP.
14. Received autologous or allogeneic cell therapy within 4 weeks, such as donor lymphocyte infusion.
15. Received autologous or allogeneic gene modified adoptive cell therapy (e.g. CAR-T, TCR-T, CAR-NK cell therapy, etc).
16. Subject received anti-tumour treatment (chemotherapy, monoclonal antibody, or hormone) within one week of screening (hydroxycarbamide is permitted until lymphodepletion).
17. Has a known history of prior malignancy, except for;

17.a. Malignancies that were treated curatively and have not recurred within 2 years prior to study treatment 17.b. Completely resected basal cell and squamous cell skin cancers 17.c. Any malignancy considered to be indolent and that has never required therapy 17.d. Completely resected carcinoma in situ of any type

18. Pregnant or lactating women.

19. Hypersensitivity to iron-dextran or murine antibodies.

20. Patients who are active participants in other interventional clinical trials at the same time. Co-enrolment is permitted for non-interventional studies if approved by the CI.

21. The Investigator believes that there are other factors that are not suitable for inclusion or influence the patient's participation or completion of the study.

22. Considered unsuitable for further intensive therapy or expected to survive less than 3 months with conventional available treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Reduction in myeloblast levels in response to TCB008 dosing | The total duration of study participation for each patient (from screening through end of study visit) is anticipated to be approximately 15 months).
  Reduction in myeloblast levels compared to baseline, measured according to the ELN AML 2022 Response Criteria.
Patient relapse and subsequent response to repeat TCB008 dosing | The total duration of study participation for each patient (from screening through end of study visit) is anticipated to be approximately 15 months).
  Measured by the numbers of patients who, after initial response, subsequently relapse and then respond to an additional infusion.
Overall response rate to TCB008 dosing | The total duration of study participation for each patient (from screening through end of study visit) is anticipated to be approximately 15 months).
  Overall response rate, defined as morphological CR, CRi, Rh, PR, and MLFS at 28-days post-infusion, measured according to the ELN AML 2022 Response Criteria.
Measurable Residual Disease in response to TCB008 dosing | The total duration of study participation for each patient (from screening through end of study visit) is anticipated to be approximately 15 months).
  MRD-negative remission (CR without MRD or CR MRD-) by multiparameter flow cytometry-based MRD (MFC-MRD) or molecular MRD (Mol-MRD) assessed by qPCR, according to the ELN AML 2022 Response Criteria.

SECONDARY OUTCOMES:
Severity of adverse events in response to TCB008 dosing | The total duration of study participation for each patient (from screening through end of study visit) is anticipated to be approximately 15 months).
  Safety assessment of AEs graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Incidence and severity of CRS and neurotoxicity in response to TCB008 dosing | The total duration of study participation for each patient (from screening through end of study visit) is anticipated to be approximately 15 months).
  Incidence and severity of cytokine release syndrome (CRS) and neurotoxicity, using the ASTCT consensus grading system.
Overall survival rates following TCB008 dosing | The total duration of study participation for each patient (from screening through end of study visit) is anticipated to be approximately 15 months).
  Overall survival assessed at 52 weeks according to the ELN AML 2022 Response Criteria.
Relapse-free survival following TCB008 dosing | The total duration of study participation for each patient (from screening through end of study visit) is anticipated to be approximately 15 months).
  Relapse-free survival assessed at 52 weeks according to the ELN AML 2022 Response Criteria.
Event-free survival following TCB008 dosing | The total duration of study participation for each patient (from screening through end of study visit) is anticipated to be approximately 15 months).
  Event-free survival assessed at 52 weeks according to the ELN AML 2022 Response Criteria.
Cumulative incidence of relapse following TCB008 dosing | The total duration of study participation for each patient (from screening through end of study visit) is anticipated to be approximately 15 months).
  Cumulative incidence of relapse assessed at 52 weeks according to the ELN AML 2022 Response Criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Nicholson, MD, Principal Investigator — Royal Marsden Hospital London
Locations (6):
- United Kingdom (6):
  - Bristol and Weston NHS foundation trust, Bristol
  - Cardiff and Vale University LHB, Cardiff
  - Queen Elizabeth University Hospital, Glasgow
  - Guys&St Thomas NHS foundation Trust, London
  - Kings College Hospital, London
  - Royal Marsden Hospital, London

IPD SHARING:
Plan to Share IPD: Undecided